CLINICAL TRIAL: NCT01407055
Title: Clinical Applications of Placebo Research: Optimizing Expectation Effects in Cardiac Surgery Patients
Brief Title: Optimizing Expectations in Cardiac Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr. Winfried Rief, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFG RI574/21-1
Record Dates: First submitted 2011-07-25; First posted 2011-08-01 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Bypass Graft Surgery (CABG); Patients' Expectations; Coronary Heart Disease
Keywords: Coronary Artery Bypass Graft Surgery (CABG); Patients' Expectations; Coronary Heart Disease; Illness Perception Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Coronary Disease | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Medical Care (No Intervention): Patients receive standard treatment protocol for Coronary Artery Bypass Graft Surgery
- Attention Control Group (Active Comparator): In addition to standard medical care patients receive a comparable amount of therapist´s attention (common and unspecific factors = supportive therapy) to the intervention group, without targeting patients' expectations.
  Interventions: Behavioral: Supportive Therapy
- Expectation Manipulation Intervention (Experimental): In addition to standard medical care patients' expectations prior to surgery are targeted in a brief psycho-educational intervention.
  Interventions: Behavioral: Expectation Manipulation Intervention

INTERVENTIONS:
Behavioral: Expectation Manipulation Intervention — The Expectation Manipulation Intervention targets patients' expectations prior to surgery (2 individual sessions, 2 phone calls). Main goal is to enhance positive outcome expectancies, as well as to improve patients' control expectations about possible side effects of the surgery and about their personal management of their coronary heart disease. Further EMI tries to correct dysfunctional beliefs about the coronary heart disease and tries to minimize fears about expected negative consequences.
  Arms: Expectation Manipulation Intervention
Behavioral: Supportive Therapy — Supportive therapy employs common factors such as elicitation of affect, reflective listening, feeling understood, but provides no explicit theoretical formulation to the patient. Supportive therapy thus provides a control condition for common factors and therapist attention but lacks the specific intervention part. It will be delivered in the same frequency and at the same time points as the Expectation Manipulation Intervention (2 individual sessions, 2 phone calls).
  Arms: Attention Control Group

SUMMARY:
The purpose of this study is to evaluate the potential benefit of targeting patients' expectations before coronary artery bypass graft surgery through a brief psychoeducational intervention.

DETAILED DESCRIPTION:
Coronary artery bypass graft surgery (CABG) is an extremely invasive medical intervention.It is postulated that even under these conditions, treatment outcome is substantially determined by non-specific effects, e.g. patient's expectation. Targeting patients' expectations at an early stage might have potential to optimize outcomes after cardiac surgery. The purpose of this research project is to optimize patients' outcome expectations before undergoing cardiac surgery through a brief psycho-educational program. Using a randomized controlled design, 180 patients who are scheduled to undergo elective CABG are randomly assigned either to standard medical information alone, or to an additional expectation manipulation intervention (EMI) during the two weeks before surgery, or to an attention-control group ("supportive therapy"). The main goal is to enhance positive expectations (surgery 'non-specific effects') about favorable outcome through EMI, about coping abilities to deal with adverse events, and to reduce negative expectations and misconceptions. Assessment takes place before and after EMI, 10 days after surgery and 6 months later; same assessment points are used for the 2 control conditions. Primary outcome is disability, which has been shown to be strongly determined by patient's expectation in previous studies. Moreover, psychological and biological predictors and mediators of treatment success are analyzed. A positive result for this expectation intervention would have major implications for clinical practice. In order to optimize treatment outcome, it is not only necessary to improve the treatment-specific procedures (e.g., cardiac surgery) but also to address non-specific factors such as patients' expectations.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled on the elective waiting list for first time coronary artery bypass graft surgery wiht the use of heart-lung-apparatus at the Department of Cardiovascular Surgery, Medical School, University of Marburg
* Sufficient knowledge of German language
* Ability to give informed consent

Exclusion Criteria:

* Emergency surgery
* Presence of a serious comorbid psychiatric condition
* Presence of a life threatening comorbid medical condition
* Current participation in other research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Disability 6 months after surgery, controlled for baseline disability (Pain Disability Index; PDI) | 6 months after surgery

SECONDARY OUTCOMES:
Change in Patients' Expectations from Baseline/Pre-Intervention (expected average of 10 days before surgery) to hospital admission/Post-Intervention (expected average of 1 day before surgery). | From 10 days before surgery untill 1 day before surgery
  Prospective Illness Perception 6 months after surgery (Expected Illness Perception Questionnaire; IPQ-E), Positive Health Expectation Scale (PHES), Expected Disability (PDI-E)
Change in Cardiac Anxiety (Cardiac Anxiety Questionnaire; CAQ) from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery
Change in Physical Activity (International Physical Activity Questionnaire; IPAQ) from Baseline (an expected average of 10 days before surgery) to 6 months after surgery. | From 10 days before surgery to 6 months after surgery
Change in Health Related Quality of Life (SF-12) from Baseline (expected average of 10 days before surgery) to 6 months after surgery. | From 10 days before surgery to 6 months after surgery
Change in physical symptoms, subjective side effects and post-surgery complaints (Generic Assessment of Side Effects Scale; GASE-P)from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery
Change in Hospital Anxiety and Depression Scale (HADS)from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery.
Change in Beliefs about Medications (Beliefs about Medications Questionaire; BMQ)from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery.
Change in Working ability from Baseline (expected average of 10 days before surgery) to 6 months after surgery. | From 10 days before surgery to 6 months after surgery.
Satisfaction wiht the intervention. | Expected average of 1 day before surgery (but after the intervention).
Cardiothoracic surgeons' rating of the surgery success | Expected average of 1 day after surgery
Additional treatments during follow-up | 6 months after surgery
  Additional Treatments, rehospitalizations, cardiac sport groups, rehabilitations programms, etc.
Blinded Expert Rating of medical and psychological status at follow-up | 6 months after surgery
Change in Sleep Quality from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery.
Change in neuroendocrine and immunological measures from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery.
  cortisol, inflammatory processes, catecholamines
Patient Pre-/Peri-/Postoperative Health Status retrospectively collected from patient file | 6 months after surgery
  From Patient file:
  Left ventricular ejection fraction (EF), Body Mass Index, Blood pressure, Smoking status, Cardiac Operative Risk (EuroSCORE), New York Heart Association classification (NYHA), Canadian Cardiovascular Society grading of angina pectoris (CCS), Number of diseased coronary vessels, Previous myocardial infarctions, extra-cardiac arteriopathy, non-cardiac comorbidities, surgery procedure, surgery complications and in-hospital post surgery complications, time spent on the intensive care unit, inpatient days until discharge
Patients' experience with prior surgeries | Baseline (expected average of 10 days before surgery)
  Rating of experience with own prior surgeries. Rating of experience with surgeries of close others.
Enriched Social Support Inventory | Baseline (expected average 10 days before surgery)
Occurrence of major life events since surgery | 6 months after surgery
Change in Patients' Illness Perception (Brief Illness Perception Questionnaire (B-IPQ) from 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery. | From 10 days before surgery to 1 day before surgery to 10 days after surgery to 6 months after surgery
Satisfaction with the intervention | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Department of Clinical Psychology and Psychothearpy, Philipps University of Marburg; Rainer Moosdorf, Prof. Dr., Principal Investigator — Department of Cardiac and Thoracic Vessel Surgery, Heart Centre, Philipps University of Marburg
Locations (1):
- Philipps University of Marburg, Marburg, Hesse, Germany

REFERENCES:
- [Background] Laferton JA, Shedden Mora M, Auer CJ, Moosdorf R, Rief W. Enhancing the efficacy of heart surgery by optimizing patients' preoperative expectations: study protocol of a randomized controlled trial. Am Heart J. 2013 Jan;165(1):1-7. doi: 10.1016/j.ahj.2012.10.007. Epub 2012 Nov 14. PMID 23237127
- [Derived] Horn N, Laferton JAC, Shedden-Mora MC, Moosdorf R, Rief W, Salzmann S. Baseline depressive symptoms, personal control, and concern moderate the effects of preoperative psychological interventions: the randomized controlled PSY-HEART trial. J Behav Med. 2022 Jun;45(3):350-365. doi: 10.1007/s10865-022-00319-0. Epub 2022 May 6. PMID 35522399
- [Derived] Salzmann S, Euteneuer F, Laferton JAC, Shedden-Mora MC, Schedlowski M, Moosdorf R, Rief W. IL-8 and CRP moderate the effects of preoperative psychological interventions on postoperative long-term outcomes 6 months after CABG surgery - The randomized controlled PSY-HEART trial. Brain Behav Immun. 2021 Jan;91:202-211. doi: 10.1016/j.bbi.2020.09.028. Epub 2020 Sep 28. PMID 33002633
- [Derived] Salzmann S, Euteneuer F, Laferton JAC, Auer CJ, Shedden-Mora MC, Schedlowski M, Moosdorf R, Rief W. Effects of Preoperative Psychological Interventions on Catecholamine and Cortisol Levels After Surgery in Coronary Artery Bypass Graft Patients: The Randomized Controlled PSY-HEART Trial. Psychosom Med. 2017 Sep;79(7):806-814. doi: 10.1097/PSY.0000000000000483. PMID 28846584
- [Derived] Auer CJ, Laferton JAC, Shedden-Mora MC, Salzmann S, Moosdorf R, Rief W. Optimizing preoperative expectations leads to a shorter length of hospital stay in CABG patients: Further results of the randomized controlled PSY-HEART trial. J Psychosom Res. 2017 Jun;97:82-89. doi: 10.1016/j.jpsychores.2017.04.008. Epub 2017 Apr 19. PMID 28606503
- [Derived] Rief W, Shedden-Mora MC, Laferton JA, Auer C, Petrie KJ, Salzmann S, Schedlowski M, Moosdorf R. Preoperative optimization of patient expectations improves long-term outcome in heart surgery patients: results of the randomized controlled PSY-HEART trial. BMC Med. 2017 Jan 10;15(1):4. doi: 10.1186/s12916-016-0767-3. PMID 28069021
- See also: Homepage of the transregional DFG research unit FOR 1328: Expectation and conditioning as basic processes of the placebo and nocebo response: From neurobiology to clinical applications — http://placeboforschung.de/